CLINICAL TRIAL: NCT01859091
Title: Pilot Study to Evaluate Non-Invasive Subcutaneous Fat Reduction in the Submental Area Using Cryolipolysis
Brief Title: Pilot Study on the Submental Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA13-004
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fat Reduction (Experimental)
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of cryolipolysis for non-invasive reduction of submental fat.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Presence of submental fat, which in the investigator's opinion, may benefit from the treatment.
3. No weight change exceeding 10 pounds in the preceding month.
4. Agreement to maintain his/her weight (i.e., within 10 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
5. Subject has signed a written informed consent form.

Exclusion Criteria

1. Skin laxity in the neck or chin area for which reduction in submental fat may.
2. Evidence of any cause of enlargement in the submental area other than localized subcutaneous fat.
3. Enlargement on the anterior neck that may prevent the proper placement of the applicator.
4. Treatment with dermal fillers, radiofrequency or laser procedures, or chemical peels in the neck or chin area.
5. Botulinum toxin injections within the neck or chin area.
6. History of a fat reduction procedure in the area of intended treatment.
7. History of prior surgery in the area of intended treatment.
8. Current dental infection.
9. Known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
10. Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
11. Impaired skin sensation or thermal sensitivity in the intended treatment area.
12. Open or infected wounds in the intended treatment area.
13. Currently taking or has taken diet pills or weight control supplements within the past month.
14. Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
15. Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
16. Pregnant or intending to become pregnant in the next 5 months.
17. Lactating or has been lactating in the past 6 months.
18. Unable or unwilling to comply with the study requirements.
19. Currently enrolled in a clinical study of any other unapproved investigational drug or device.
20. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Reduction: The Zeltiq System: Non-invasive cooling applied to the treatment area with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | Fat Reduction
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fat Reduction
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device and/or Procedure Related Adverse Events (AEs) and Device-related Serious Adverse Events (SADEs)
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not considered related to treatment. A serious adverse event (SAE) was an AE that resulted in death, serious deterioration in health, permanent impairment of a body structure/function, was life-threatening, required hospitalization or medical/surgical intervention, led to fetal distress or death, congenital abnormality, or birth defect. An ADE was any sign, symptom, or disease that was determined by the Investigator to have a causal relationship or possible causal relationship with the investigational device, including any AE resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the device or from use error or intentional misuse of the device. A SADE was an ADE that resulted in any of the consequences characteristic of an SAE.
Time Frame: 8-weeks post treatment
Population: All enrolled subjects (Fat Reduction group) who received treatment.
Measure: Number; unit: participants
Arm/Group | Fat Reduction
Number analyzed (Participants) | 14
participants
  Device and/ or Procedure Related AEs | 0
  SADEs | 0

2. Secondary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 8-week post-treatment ultrasound measurements taken in the area treated with the device, and in the adjacent untreated control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes were normalized for each subject by subtracting the change in control (untreated area) from the change in treated area to remove the influence of weight variations. Success is defined as, on average, at least a 1mm or greater reduction in fat layer thickness for the treated region as compared to the untreated control. Results indicate the mean fat layer reduction in mm.
Time Frame: Baseline, 8-weeks post treatment
Population: Per Protocol population consisted of participants who received treatment and had ultrasound data collected at the 8-weeks post treatment time point.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Fat Reduction
Number analyzed (Participants) | 13
mm | 0.5 [0.14 to 0.85]

3. Secondary Outcome: Number of Pre- and Post-Treatment Photograph Pair Reviews (Correctly Identified by an Internal Reviewer Panel of 4 Reviewers)
Description: Photographs of the treatment areas taken at baseline and 8-weeks after final treatment were assessed for visible changes in contour in the treated areas. Pre- and post-treatment photograph pairs were randomized and reviewed by a blinded reviewer panel of 4 reviewers.
Time Frame: 8-weeks post treatment
Population: Per Protocol population consisted of participants who received treatment, had a weight change of no more than 10 pounds, and did not become pregnant at the time the 8-week assessments were performed compared to the weight obtained at the first treatment visit.
Measure: Number; unit: Number of correct photo pair reviews
Units Other Than Participants: Photograph Pair Reviews
Arm/Group | Fat Reduction
Number analyzed (Participants) | 14
Number analyzed (Photograph Pair Reviews) | 56
Number of correct photo pair reviews | 23

ADVERSE EVENTS:
Time Frame: Any adverse event information was collected from the time of study enrollment through the 8-week post-treatment follow-up visit, up to 10 weeks.
Description: The Safety Population consisted of all enrolled participants who received at least one study treatment.
Arm/Group | Fat Reduction
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No